CLINICAL TRIAL: NCT03466762
Title: Resilience and Quality of Life of Head & Neck Cancer and Brain Tumor Survivors in Pakistan
Brief Title: Resilience and Quality of Life Among Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Nida Zahid, Senior Instructor Research, Aga Khan University
Other Study IDs: 5154-Sur-ERC-17
Record Dates: First submitted 2018-03-01; First posted 2018-03-15 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Mental Health Wellness 1
Keywords: Quality of life; Resilience; Cancer Survivors; Life Satisfaction; Post-Cancer Depression; Coping
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non applicable — Non applicable

SUMMARY:
The main aim of this study is to evaluate the impact of head & neck cancer and brain tumors on lives of patients in Pakistan. To the best of the investigators knowledge this will be the first in-depth study to evaluate resilience and quality of life (QoL) among this group of patients. These patients encounter challenges as they battle to maintain optimistic outlook towards life. Resilience and QoL among them changes over time and may be modifiable towards increased well-being. Resilience and QoL are critical components during diagnosis, treatment, survivorship, and at the end of life. Hence, these are important traits for promoting positive psychological well-being. Through this study the investigators will be able to identify problems faced by such patients in our setting. the investigators will be able to plan appropriate interventions to improve a person's resiliency and quality of life, reduce depression and anxiety, and increase their satisfaction with life. This study is also aimed to inform healthcare providers and researchers regarding protective or risk characteristics for coping with cancer. Practices and resilience interventions may improve well-being and adherence to care guidelines.

The objectives of our study are:

Primary Objectives:

* To determine resilience and quality of life scores after treatment separately for head & neck cancer and Brain tumor patients in Pakistan.
* To evaluate important factors associated with resilience and quality of life after treatment separately for head & neck cancer and Brain tumor patients in Pakistan.

Secondary Objective:

• To examine the relationship between resilience and quality of life after treatment separately for head & neck cancer and Brain tumor patients in Pakistan.

It will be an analytical cross sectional study design. The study will be conducted at the Aga Khan University Hospital, Karachi. Study participants will be men and women greater than 18 years, with brain tumors or head & neck cancer fulfilling the eligibility criteria. Approximately 250 patients will be recruiting with brain tumors and 250 with head & neck cancer. Validated tools will be used to measure resilience and QoL.

DETAILED DESCRIPTION:
Background In 2012, around 14.1 million new cases of cancer were diagnosed worldwide and another 8.2 million died from cancer. It is estimated that by 2030, these figures could increase to an alarming 26.4 million new cases and 17 million cancer-related deaths. Nearly 56% of the new cancer cases and 64% of the cancer-related deaths occur in low and middle income countries (LMICs), where there is a lack of universally available, affordable, and sustainable health care. Head and neck cancers are among the most common cancers worldwide with nearly 600,000 new cases and 300,000 deaths occurring globally every year. Brain tumors are responsible for approximately 2% of all cancer deaths. The overall incidence of brain tumors is 4-5/100,000 population per year. Cancer's diagnosis considerably affects patient's emotional and psychological status. The cancer survivors encounter various challenges, as they battle to maintain an optimistic outlook towards life. Resilience enables individuals to thrive in the face of adversity and it is believed that resilience plays an important role in a cancer survivor's life to cope with their illness, to overcome depression and improve their Health- related quality of life (HR-QoL). HR-QoL and its assessment have become increasingly important in health care, especially in the field of chronic diseases recently. HR-QoL generally refers to patients' perceptions of the effects of disease on life. It has two fundamental premises; first, a multi-dimensional concept incorporating physical, psychological, social, and emotional functional domains. Second is subjective and must be self-reported, according to the patients' own experiences. Conventionally, the endpoints of medical care for cancer patients had focused on survival rate, local control rate, or complication rate. However, assessments have lacked knowledge and understanding of the patient's mental and emotional wellbeing. Recently, resilience in the course of cancer treatment has been given immense attention. Several studies from different parts of the world on cancer survivors suggest that resilience is a protective factor for distress. A study reported resilience was likely to mediate the adverse relationship between cancer symptoms, distress and QoL for cancer survivors, indicating, resilience might play an essential role in protecting against adverse effects of cancer symptoms on QoL. It is identified, that resilience as an important changeable path can improve hope and QoL. Therefore, it is important that before initiating treatment, patients should be referred to a mental health professional for psychological/psychiatric evaluation. Resilience and QoL is a critical component during diagnosis, treatment, survivorship, and at the end of life. Hence, these are important traits for promoting positive psycho-social well-being. Resilience and QoL changes over time and may be modifiable towards increased well-being. To the best of the investigators knowledge, this will be the first in-depth study to evaluate resilience and quality of life among head & neck cancer and brain tumor patients in Pakistan. Moreover, through this study the investigators will be able to identify problems faced by such patients in their setting, enabling the investigators in the future to design interventions to improve resilience and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Individual aged > 18 years both gender
2. Had received treatment at AKUH for head & neck cancer and/or brain tumor.
3. Pakistani national currently living in Pakistan.

Exclusion Criteria

1. Known cases of any physical and/or psychiatric illness (manic disorder, schizophrenia etc.) confirmed by medical records will be excluded from the study as they may be on medications, hence we may not get the true results.
2. Patients on anti-depressants prescribed by a psychiatrist.
3. Participant with terminal disease like renal failure and stroke will be excluded because these diseases also have profound effect on quality of life and resilience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women greater than 18 years, who have received treatment for brain tumor and head & neck cancer, fulfilling the below eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Resilience of head and neck cancer and Brain tumor survivors | April 2018-March 2019
  Resilience will be measured by Wagnild & Young's 14 Item A high score represents better resilience. The respondent's choice ranges from 1 (Strongly Disagree) to 7 (Strongly Agree). The scale uses total scores rather than scores of individual items.

SECONDARY OUTCOMES:
Quality of life of head and neck cancer and Brain tumor survivors | April 2018-March 2019
  Quality of life will be measured by European Organization of Research and Treatment Of Cancer tool general (EORTC QLQ-C30) AND European Organization of Research and Treatment Of head and Neck cancer (EORTC QLQ-H&N35) AND European Organization of Research and Treatment Of Brain tumor ( EORTC QLQ-BN20) All of the scales and single-item measures scores range from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zahid N, Khalid W, Ahmad K, Bhamani SS, Azam I, Asad N, Jabbar AA, Khan M, Enam A. Resilience and quality of life (QoL) of head and neck cancer and brain tumour survivors in Pakistan: an analytical cross-sectional study protocol. BMJ Open. 2019 Sep 20;9(9):e029084. doi: 10.1136/bmjopen-2019-029084. PMID 31542743